CLINICAL TRIAL: NCT02562066
Title: A Phase 3, Double-blind, Outpatient Crossover Study to Evaluate the Efficacy and Safety of Amifampridine Phosphate (3,4 Diaminopyridine Phosphate) in Patients With Congenital Myasthenic Syndromes (CMS)
Brief Title: Amifampridine Phosphate for the Treatment of Congenital Myasthenic Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMS-001
Expanded Access: NCT02189720 (Approved for marketing)
Record Dates: First submitted 2015-09-24; First posted 2015-09-29 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-02

CONDITIONS: Myasthenic Syndromes, Congenital
MeSH Terms: conditions — Myasthenic Syndromes, Congenital | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- amifampridine phosphate -placebo (Experimental): Each patient will participate in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate is achieved for 7 days. After this phase, half of the subjects will be randomized to receive amifampridine in Period I and then crossed over to receive placebo in Period II. Each randomized treatment period is 7 days in duration and is separated by a re-stabilization period of approximately two weeks where the subject will be returned to the stable dose administered at the end of the open-label run-in period. Dosing will be between 20 - 80 mg per day and frequency will be between 2-4 times per day.
  Interventions: Drug: amifampridine phosphate; Drug: Placebo
- placebo - amifampridine phosphate (Experimental): Each patient will participate in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate is achieved for 7 days. After this phase, half of the subjects will be randomized to receive placebo in Period I and then crossed over to receive amifampridine in Period II. Each randomized treatment period is 7 days in duration and separated by a re-stabilization period of approximately two weeks where the subject will be returned to the stable dose administered at the end of the open-label run-in period. Dosing will be between 20 - 80 mg per day and frequency will be between 2-4 times per day.
  Interventions: Drug: amifampridine phosphate; Drug: Placebo

INTERVENTIONS:
Drug: amifampridine phosphate — Amifampridine phosphate tablets 10 mg will be provided in round, white-scored tablets, and containing amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
  Other Names: 3,4 diaminopyridine phosphate, Firdapse™
Drug: Placebo — A placebo equivalent will be provided as tablets indistinguishable from the amifampridine phosphate tablets. The placebo will be administered consistent with the dose regimen of amifampridine phosphate.

SUMMARY:
This randomized, double-blind, controlled, outpatient two-period, two-treatment crossover study is designed to evaluate the efficacy and safety of amifampridine phosphate in patients (ages 2 and above) diagnosed with certain genetic subtypes of CMS and demonstrated open label (amifampridine phosphate) or history of sustained amifampridine benefit from treatment.

DETAILED DESCRIPTION:
Each patient will participate in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate is achieved for 7 days. After this phase, blinded treatment effect will be assessed in a randomized fashion of continuation or cessation of drug (Placebo) starting with Period I (duration 7 days). Following experimental Period 1, patients will be returned to the stable dose administered at the end of the open-label run-in period for approximately 2 weeks, followed by cross over treatment in Period 2 dosing for 7 days. After completion of Period 2, patients will be eligible for expanded access with restoration of open-label amifampridine phosphate at the same dose and frequency as established in the run in phase of the study.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate in this study must meet all of the following inclusion criteria:

1. Patient's or parent willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures, or the patient's legal guardian or caregiver with durable power of attorney can provide written informed consent. An assent form must also be signed if in the judgement of the IRB the children are capable of providing assent.
2. Male or female age 2 and above.
3. Body weight ≥10 kg.
4. Genetically-confirmed CMS involving acetylcholine receptor defect, Rapsyn deficiency, MuSK deficiency, Dok-7 deficiency, SYT2 deficiency,SNAP25B deficiency, and fast channel syndrome.
5. MFM 20 or 32 score equal or less than 48 or 76, respectively, at Screening.
6. In patients naïve to 3,4-DAP or amifampridine phosphate, improvement of >20% in MFM20 or MFM32 scores after open label period of up titration of dose
7. In patients previously stabilized on 3,4-DAP or amifampridine phosphate, history of meaningful improvement in motor function (in opinion of investigator)
8. Willingness of patients receiving pyridostigmine, prednisone, albuterol, ephedrine, or fluoxetine to remain on a stable dose of these medications throughout the study interval.
9. Female patients of childbearing potential must have a negative pregnancy test (serum human chorionic gonadotropin [HCG] at Screening); and must practice effective, reliable contraceptive regimen during the study.
10. Ability to participate in the study based on overall health of the patient and disease prognosis, as applicable, in the opinion of the investigator; and able to comply with all requirements of the protocol.

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria are not eligible to participate in the study:

1. CMS subtype diagnosis of acetylcholinesterase deficiency, slow-channel syndrome, LRP4 deficiency, and plectin deficiency.
2. Cardiac conduction defects on Screening ECG.
3. Seizure disorder.
4. Abnormal liver function tests at Screening.
5. Abnormal kidney function tests at Screening.
6. Abnormal electrolyte values at Screening.
7. Pregnancy or breastfeeding at Screening or planning to become pregnant at any time during the study.
8. Any systemic bacterial or other infection, which is clinically significant in the opinion of the investigator and has not been treated with appropriate antibiotics.
9. Treatment with an investigational drug (other than amifampridine phosphate), device, or biological agent within 30 days before Screening or while participating in this study.
10. Any other medical condition that, in the opinion of the investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confound the assessment of the patient.
11. History of drug allergy to any pyridine-containing substances or any amifampridine phosphate excipient(s).

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2019-08 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Crawford, M.D., Principal Investigator — Johns Hopkins Pediatric Neurology
Locations (4):
- United States (4):
  - UCLA Department of Neurology, Los Angeles, California
  - Johns Hopkins Pediatric Neurology, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 08 February 2016 - 24 January 2019 and was conducted at six sites in the United States and two sites in Canada, although one site (Montreal Neurological Institute and Hospital) did not enroll any patients.
Pre-assignment Details: Screening ensured patients met I/E criteria. Patients naïve to amifampridine began open-label titration until a stable dose and frequency was achieved for 7 days. Demonstrated efficacy (assessed by improvement on the MFM) was required to participate in the randomized portion of the study. Patients already on a stable dose with hostory of meaningful improvement were eligible immediately and transitioned to an equivalent dose of amifampridine phosphate for 7 days prior to randomization.
Groups:
- Amifampridine Phosphate - Placebo: Each patient will participate in an open-label unblinded drug escalation/treatment run-in phase for up to 4 weeks until stable dose and frequency of amifampridine phosphate is achieved for 7 days. After this phase, half of the subjects will be randomized to receive amifampridine in Period I and then crossed over to receive placebo in Period II. Each randomized treatment period is 7 days in duration and is separated by a re-stabilization period of approximately two weeks where the subject will be returned to the stable dose administered at the end of the open-label run-in period. Dosing will be between 20 - 80 mg per day and frequency will be between 2-4 times per day.
  Amifampridine Phosphate: Amifampridine phosphate tablets 10 mg will be provided in round, white-scored tablets, and containing amifampridine phosphate formulated to be the equivalent of 10 mg amifampridine base per tablet.
  Placebo: A placebo equivalent will be provided as tablets indistinguishable from the amifampridine phosphate tablets. The placebo will be administered consistent with the dose regimen of amifampridine phosphate.
- Amifampridine Phosphate Only: Patients receiving amifampridine during the open-label run-in period but were not randomized for the crossover portion of the study.
Period: Overall Study
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate | Amifampridine Phosphate Only
Started | 8 | 8 | 4
Completed | 7 | 7 | 0
Not Completed | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized patients who have received at least one dose of study medication. Note that subjects in the Amifampridine Phosphate Only arm are excluded from this analysis, as they were not randomized for inclusion in the crossover portion of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 | 12
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.59 (15.70) | 27.35 (25.00) | 19.97 (21.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Subject Global Impression (SGI) Score Summary: Mann-Whitney Main Effects Test Results; SGI Score Mixed Model Analysis
Description: Subject Global Impression (SGI) rates the subject's impression of the effects of the study medication during the preceding week with max score =7 (most satisfied) and min score =1 (least satisfied). It will be completed at D0 (baseline for Study Period 1), D8, D21 (baseline for Study Period 2), and D29. Change from baseline (CFB) will be assessed for Study Period 1 (difference in SGI score from D0 to D8), Study Period 2 (difference in SGI score from D21 to D29) and the change in CFB from Study Period 1 to Study Period 2 (difference between CFB during Study Period 1 and CFB during Study Period 2). A Mann-Whitney-Wilcoxon test for equality of the CFB results in the two treatments in Period 1 and for the equality of the CFB results in the two treatment sequences will be conducted. A mixed effects liner model will be fit with the SGI raw scores as a response and study arm, treatment, period, age group and mutation type as fixed effect terms and patient as a random effect.
Time Frame: Study Period 1: Baseline (Day 0), Day 8; Study Period 2: Baseline (Day 21), Day 29
Population: The Full Analysis Set consists of all randomized patients who receive at least one dose of study medication and have at least one post-treatment efficacy assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate
Number analyzed (Participants) | 8 | 8
Scores on a scale
  Study Period 1: CFB in SGI Score at Day 8 | -0.13 (1.81) | -1.75 (2.12)
  Study Period 2 : CFB in SGI Score at Day 29 | -0.75 (1.75) | -1.14 (1.68)
Statistical Analysis 1: Comparison: Amifampridine Phosphate - Placebo vs Placebo - Amifampridine Phosphate; A Mann-Whitney-Wilcoxon test for equality of the change from baseline (CFB) in the two treatments in Period 1 will be presented; Test type: Other; p = 0.085, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.63 — Results show the difference in mean CFB at the end of Study Period 1
Statistical Analysis 2: Comparison: Amifampridine Phosphate - Placebo; A mixed effects linear model will be fit to the data with SGI raw scores as the response and fixed effect terms for treatment, period, age group, mutation type and sequence*period, and a random effect for patient. The LSMeans for the estimated difference between treatments in Period 1 along with a 95% confidence interval for this difference; Test type: Other; Mixed Models Analysis; Mean Difference (Net) = 0.56, 95% CI 2-sided [-0.97 to 2.09] — Results show the LSMeans for the estimated difference between treatments in Period 1 along with a 95% confidence interval for this difference

2. Secondary Outcome: Motor Function Measure 32 (MFM-32) Score Summary: Mann-Whitney Main Effect Test Results, MFM-32 Score Mixed Model Analysis
Description: Motor Function Measure 32 (MFM-32) evaluates the severity and progression of motor function in patients 7 years of age or older with max total score = 96 (best score) and min total score =0 (worst score). It will be completed at D0 (baseline for Study Period 1), D8, D21 (baseline for Study Period 2) and D29. CFB will be assessed for Study Period 1 (difference in MFM-32 from D0 to D8), Study Period 2 (difference in MFM-32 from D21 to D28) and the change in CFB from Study Period 1 to Study Period 2 (difference between CFB during Study Period 1 and CFB during Study Period 2). A Mann-Whitney-Wilcoxon test for equality of CFB results in the two treatments in Period 1 and for the equality of the CFB results in the two treatment sequences will be conducted. A mixed effects linear model will be fit to the overall MFM-32 score as the response variable and fixed effect terms for treatment, period, age group, genetic mutation type, and sequence*period and a random effect for patient.
Time Frame: Study Period 1: Baseline (Day 0), Day 8; Study Period 2: Baseline (Day 21), Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate
Number analyzed (Participants) | 8 | 8
Score on a Scale
  Study Period 1: CFB in Overall MFM-32 Score at Day 8: number analyzed (Participants) | 4 | 6
  Study Period 1: CFB in Overall MFM-32 Score at Day 8 | 3.00 (3.92) | -0.17 (4.58)
  Study Period 2: CFB in Overall MFM-32 Score at Day 29: number analyzed (Participants) | 4 | 5
  Study Period 2: CFB in Overall MFM-32 Score at Day 29 | 0.75 (2.22) | -0.60 (0.89)
Statistical Analysis 1: Comparison: Amifampridine Phosphate - Placebo vs Placebo - Amifampridine Phosphate; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.376, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 3.17 — Results show the difference in mean CFB at the end of Study Period 1
Statistical Analysis 2: Comparison: Amifampridine Phosphate - Placebo vs Placebo - Amifampridine Phosphate; A mixed effects linear model will be fit to the data with Overall MFM-32 scores as the response and fixed effect terms for treatment, period, age group, mutation type and sequence*period, and a random effect for patient. The LSMeans for the estimated difference between treatments in Period 1 along with a 95% confidence interval for this difference; Test type: Other; Mixed Models Analysis; Mean Difference (Net) = 1.14, 95% CI 2-sided [-2.31 to 4.58] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Motor Function Measure 20 (MFM-20) Score Mixed Model Analysis, MFM-20 Score Mixed Model Analysis
Description: Motor Function Measure 20 (MFM-20) evaluates the severity and progression of motor function in patients 2 to 6 years of age with max total score = 60 (best score) and min total score =0 (worst score). It will be completed at D0 (baseline for Study Period 1), D8, D21 (baseline for Study Period 2) and D29. CFB will be assessed for Study Period 1 (difference in MFM-20 from D0 to D8), Study Period 2 (difference in MFM-20 from D21 to D28) and the change in CFB from Study Period 1 to Study Period 2 (difference between CFB during Study Period 1 and CFB during Study Period 2). A Mann-Whitney-Wilcoxon test for equality of CFB results in the two treatments in Period 1 and for the equality of the CFB results in the two treatment sequences will be conducted. A mixed effects linear model will be fit to the overall MFM-32 score as the response variable and fixed effect terms for treatment, period, age group, genetic mutation type, and sequence*period and a random effect for patient.
Time Frame: Study Period 1: Baseline (Day 0), Day 8; Study Period 2: Baseline (Day 21), Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Amifampridine Phosphate - Placebo | Placebo - Amifampridine Phosphate
Number analyzed (Participants) | 8 | 8
Score on a Scale
  Study Period 1: CFB in Overall MFM-20 Score at Day 8: number analyzed (Participants) | 4 | 2
  Study Period 1: CFB in Overall MFM-20 Score at Day 8 | -1.50 (4.20) | -0.50 (6.36)
  Study Period 2: CFB in Overall MFM-20 Score at Day 29: number analyzed (Participants) | 4 | 2
  Study Period 2: CFB in Overall MFM-20 Score at Day 29 | -0.75 (0.50) | 1.50 (2.12)
Statistical Analysis 1: Comparison: Amifampridine Phosphate - Placebo vs Placebo - Amifampridine Phosphate; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.800, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -1.00 — Results show the difference in mean CFB at the end of Study Period 1
Statistical Analysis 2: Comparison: Amifampridine Phosphate - Placebo vs Placebo - Amifampridine Phosphate; A mixed effects linear model will be fit to the data with Overall MFM-20 scores as the response and fixed effect terms for treatment, period, age group, mutation type and sequence*period, and a random effect for patient. The LSMeans for the estimated difference between treatments in Period 1 along with a 95% confidence interval for this difference; Test type: Other; Mixed Models Analysis; Mean Difference (Net) = 0.63, 95% CI 2-sided [-5.25 to 6.50] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were recorded for each patient from the time informed consent was obtained and continues through four weeks after the last dose or at the early discontinuation visit, for a total of approximately 14 weeks. Non-serious AEs were recorded for each patient after informed consent is obtained and the first administration of study drug (on Day 1 of run-in) through the last visit or at the early discontinuation visit, for a total of approximately 10 weeks .
Groups:
- Amifampridine Phosphate: Treatment administered to the patient at the time of onset of the AE. Includes patients who received amifampridine phosphate during the run-in period who were not randomized for inclusion in the crossover portion of the study.
- Placebo: Treatment administered to the patient at the time of onset of the AE.
Arm/Group | Amifampridine Phosphate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 11/20 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amifampridine Phosphate (N=20) | Placebo (N=20)
Pyrexia (General disorders) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amifampridine Phosphate (N=20) | Placebo (N=20)
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 1 | 0
Allergy to animal (Immune system disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anger (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT02562066/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02562066/SAP_001.pdf